CLINICAL TRIAL: NCT05572749
Title: Double-blind Randomized Cross-over Clinical Trial of Crocus Kozanis Administration in Obese Children and Adolescents
Brief Title: Clinical Trial of Crocus Kozanis Administration in Obese Children and Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Assimina Galli-Tsinopoulou, Professor in Paediatrics-Paediatric Endocrinology, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Crocus Kozanis & Child Obesity
Record Dates: First submitted 2022-09-13; First posted 2022-10-10 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: PreDiabetes; Obesity; Dyslipidemias
MeSH Terms: conditions — Prediabetic State; Obesity; Dyslipidemias | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): Participants of Arm 1 are going to be administered Crocus Kozanis for 12 weeks (30mg twice per day), wash-out period for 12 weeks and metformin (1000mg once per day) for 12 weeks.
  Interventions: Dietary Supplement: Crocus Kozanis; Drug: Metformin
- Arm 2 (Experimental): Participants of Arm 2 are going to be administered metformin (1000mg once per day) for 12 weeks, wash-out period for 12 weeks and Crocus Kozanis (30mg twice per day) for 12 weeks.
  Interventions: Dietary Supplement: Crocus Kozanis; Drug: Metformin
- Arm 3 (Placebo Comparator): Participants of Arm 3 are going to be administered placebo (5ml twice per day) for 12 weeks
  Interventions: Dietary Supplement: Placebo of Crocus Kozanis

INTERVENTIONS:
Dietary Supplement: Crocus Kozanis — In this study, intervention will be the administration of Crocus Kozanis dietary supplement. Crocus Kozanis is a herb which is cultivated in Kozani, Greece.
  Other Names: Saffron; Crocus Sativus; Saffron Kozanis
  Arms: Arm 1; Arm 2
Dietary Supplement: Placebo of Crocus Kozanis — Placebo of Crocus Kozanis
  Arms: Arm 3
Drug: Metformin — Metformin will be administered in a dosage of 1000mg per day. Metformin is a formally approved therapy for children with diabetes in Europe.
  Other Names: Metformin Hydrochloride
  Arms: Arm 1; Arm 2

SUMMARY:
The study aims to investigate possible effects of per os Crocus Kozanis administration in children and adolescents with obesity

ELIGIBILITY:
Inclusion Criteria:

* Age above 10 year-old
* Diagnosis of Obesity according to International Obesity Task Force Criteria
* Presence of impaired glucose tolerance and/or impaired fasting glucose

Exclusion Criteria:

* Overt diabetes (any type)
* Diagnosis of any chronic disease
* Previous use of dietary supplement with Crocus or Crocus Sativus
* Administration of chronic medication

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Glycemic control | Glycemic control will be assessed for each participant at the beginning of the study and thereafter every 12 weeks, up to 9 months (week 0, week 12, week 24, week 36).
  Glycemic control will be assessed with glycated hemoglobin (ΗbA1c%) and/or oral glucose tolerance test (OGTT)

SECONDARY OUTCOMES:
Lipidemic profile | Lipidemic profile will be assessed for each participant at the beginning of the study and thereafter every 12 weeks, up to 9 months (week 0, week 12, week 24, week 36).
  Lipidemic profile will be assessed with levels of cholesterol, triglycerides, HDL and LDL in fasting state

CONTACTS AND LOCATIONS:
Overall Officials: Assimina Galli-Tsinopoulou, Professor, Study Director — Aristotle University Of Thessaloniki
Locations (1):
- Unit of Paediatric Endocrinology and Metabolism, 2nd Department of Paediatrics, AHEPA University Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No